CLINICAL TRIAL: NCT01174927
Title: The Effects of Diacetylmorphine (Heroin) on Human Brain Functions and Stress Response
Brief Title: Effects of Diacetylmorphine (DAM) on Brain Function and Stress Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DAM2010_01; SNF127544 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Opiate
Keywords: Substance use disorder; Stress
MeSH Terms: conditions — Substance-Related Disorders | interventions — Heroin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heroin-dependent patients_1 (Active Comparator): daily dose of diacetylmorphine (30 mg to 500 mg) in 5 ml
  Interventions: Drug: diacetylmorphine (DAM)
- Heroin-dependent patients_2 (Placebo Comparator): 5 ml saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: diacetylmorphine (DAM) — The heroin-dependent patients will administer either their individual dose of prescribed DAM dose or placebo (saline) through an indwelling intravenous line. Afterwards they will complete four experimental paradigms testing response inhibition, emotional processing and working memory while brain responses are measured with fMRI. Before and after the fMRI investigation cortisol samples, DAM blood levels, neurophysiological and psychological stress parameters, such as skin conductance, heart rate, anxiety, anger, and heroin craving will be measured.
  Other Names: heroin
  Arms: Heroin-dependent patients_1
Other: Placebo — Saline
  Arms: Heroin-dependent patients_2

SUMMARY:
The aims of the study are to investigate the effects of diacetylmorphin (heroin) on brain using functional magnetic resonance imaging (fMRI), coupled with measurements of cortisol concentrations and neurophysiological stress parameters during the presentation of emotional and cognitive stimuli in patients with heroin dependence.

DETAILED DESCRIPTION:
Background: Heroin dependence (HD) is a chronic relapsing brain disorder that is defined by a compulsion to seek and use heroin, and a loss of control in limiting intake.

The prescription of diacetylmorphine (heroin) itself for maintenance has become an established treatment in several European countries. However, the neurobiological effects of diacetylmorphine (DAM) on brain function and stress response have not been studied so far. Imaging the acute effects of DAM administration during stress stimuli would elucidate the neurocircuitry and neurobiology of substance use in patients with HD.

Working hypothesis: The investigators expect that DAM attenuates the engagement of brain regions involved in response inhibition (prefrontal and anterior cingulate cortex), emotional processing (amygdala) and working memory (frontal and mediotemporal cortex). Additionally, we hypothesize that DAM reduces stress response (cortisol, heart rate, skin conductance) to emotional and cognitive stimuli.

Methods: Thirty heroin-dependent patients on stable heroin maintenance will be examined in a randomized placebo-controlled crossover design. They will be compared with 30 heroin-dependent age- and gender-matched but otherwise healthy volunteers receiving saline. The heroin-dependent patients will administer either their individual dose of prescribed DAM dose or saline through an indwelling intravenous line. Afterwards they will complete four experimental paradigms testing response inhibition, emotional processing and working memory while brain responses are measured with fMRI. Before and after the fMRI investigation cortisol samples, DAM blood levels, neurophysiological and psychological stress parameters, such as skin conductance, heart rate, anxiety, anger, and heroin craving will be measured.

Expected value of the proposed project: DAM effects on brain function and stress will advance our understanding of the mechanisms underlying HD. It is the first neuroimaging study investigating the neural basis of HD after intravenous DAM administration in humans.

Determining the neurofunctional and neurophysiological basis of heroin dependence may facilitate clinical diagnosis and improve clinical interventions such as prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* other psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
brain functions | 1 hour

SECONDARY OUTCOMES:
stress response | pre and post stress measurements

CONTACTS AND LOCATIONS:
Overall Officials: Marc Walter, MD, Principal Investigator — UPK, University Hospital Basel
Locations (1):
- UPK, Basel, Basel, Switzerland

REFERENCES:
- See also: clinic homepage — http://www.upkbs.ch